CLINICAL TRIAL: NCT04674319
Title: Attending to External Cues and Movement Strategies in Parkinson Disease: Feasibility in Ecological Setting.
Brief Title: Attending to External Cues and Movement Strategies in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galit Yogev-Seligmann (Other)
Responsible Party: Sponsor-Investigator, Galit Yogev-Seligmann, Prinicipal Investigator, University of Haifa
Organization: University of Haifa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 052/19
Record Dates: First submitted 2020-09-01; First posted 2020-12-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Gait; Attention; External cues
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain engagement while using compesatory modes for walking (Experimental): Brain engagemnent (recruitment of attention) is measured during four walking conditions
  Interventions: Behavioral: external cues and cogntive movement strategies

INTERVENTIONS:
Behavioral: external cues and cogntive movement strategies — external cueing are sensory stimuli such as auditory (e.g. rhythmic metronome beats) or or visual (e.g. spaced lines on the floor). Cognitive movement strategies refer to focusing attention on a specific parameter of gait (e.g. step length, arm swing).
  In the study participants walk under four walking conditions:1)usuall (baseline) walking 2)walking while attending to external cues wich will be applied via metronome beats. The number of beats per minute is adjusted to each participant's steps number per minute. 3)walking with movement cognitive strategy: participants are requested to focus on their step length- and focus on increasing their step length while walking 4) Dual tasking-walking while performing a cognitive task.
  During the four walking conditions Brain engegament will be measured, using the single-channel EEG system (Brain-MARC LTD) described in the follwing outcomes measures section.

SUMMARY:
People with Parkinson's disease use compensatory strategies to overcome typical gait disturbances. These strategies rely on attentional mechanisms, however people with Parkinson disease suffer of decline in cognitive function. Therefore, the current study aims at exploring brain engagement and focus of attention process during walking with these compensatory strategies, in people with Parkinson disease. Such exploration would assist in understanding the feasibility of the compensatory strategies in daily lives of people with Parkinson's disease.

DETAILED DESCRIPTION:
External cues and cognitive movement strategies are common compensatory modes that people with Parkinson's disease can use to overcome typical gait disturbances. It is suggested that these modes utilize alternative neural pathways, bypassing the impaired basal ganglia motor circuits in the brain. In addition, both compensatory modes, in particular the movement cognitive strategies, are suggested to rely on attentional mechanisms.

Cognitive deficits are common in PwP and include among others, impairment of attention, particularly in tasks requiring internal control of attention. Considering that gait compensatory modes may rely on cognitive function, in particular the cognitive movement strategies, it is not clear whether People with Parkinson's disease can engaged with these strategies for a prolonged time or distance as in many cases required in daily living.

Therefore, the objectives of this study are 1) to test the effect of compensatory modes- external cueing and cognitive movement strategy on gait in prolonged walking. 2) to test whether people with Parkinson's disease can stay engaged and focus their attention to these compensatory modes for prolonged time. 3) to test whether subject's cognitive function is related to the ability to stay engaged with these compensatory modes. Subjects are recruited from a community physical- therapy groups for people with Parkinson's disease. Healthy older adults will be recruited from the community and will serve as a control group. Participants are invited for two separate evaluation sessions that includes: 1. Assessment of background characteristic: demographic details, severity of disease ( assessed by the Unified Parkinson's Disease Rating Scale-UPDRS), Levodopa Equivalent Dose (LED), freezing of gait questionnaire (FOG-Q) and Montreal cognitive assessment (MoCA).

2. Evaluation of gait while attending to external cues and cognitive movement strategy.

3. Evaluation of brain engagement during gait 4. Computerized cognitive assessment

ELIGIBILITY:
Inclusion Criteria for people with Parkinson's disease:

* Diagnosis of Parkinson's disease
* Age of 50-85
* Able to walk independently in daily lives.

Inclusion Criteria for the control group:

* Age of 50-85
* Able to walk independently in daily lives.

Exclusion Criteria for people with Parkinson's disease:

* Use of assistive hearing device
* Suffer of hearing impairment (by self-declaration)
* Suffer of dementia (MoCa test score above 21)
* Suffer of any orthopedic condition
* Pains or other health condition that may affect gait except of PD

Exclusion Criteria for the control group:

* Use of assistive hearing device
* Suffer of hearing impairment (by self-declaration)
* Suffer of dementia (MoCa test score above 21)
* Suffer of any orthopedic condition
* Pains or other health condition that may affect gait

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Gait speed- Physiological measurement of gait | Through study completion, an average of 1 year
  Gait speed is measured with the Mobility Lab OPAL system (APDM, USA) consisting of three small inertial measurement units (IMU sensors including 3D accelerometers and 3D gyroscopes sampled at 128 Hz, MobilityLab, APDM Inc., Portland, OR). IMUs were attached at the participant's ankles, and lumbar region using elastic Velcro straps. These sensors are measuring gait speed (meters per second).
Step length- Physiological measurement of gait | Through study completion, an average of 1 year
  Step length is measured with the Mobility Lab OPAL system (APDM, USA) consisting of three small inertial measurement units (IMU sensors including 3D accelerometers and 3D gyroscopes sampled at 128 Hz, MobilityLab, APDM Inc., Portland, OR). IMUs were attached at the participant's ankles, and lumbar region using elastic Velcro straps. These sensors are measuring step length (cm).
Cadence- Physiological measurement of gait | Through study completion, an average of 1 year
  Cadence is measured with the Mobility Lab OPAL system (APDM, USA) consisting of three small inertial measurement units (IMU sensors including 3D accelerometers and 3D gyroscopes sampled at 128 Hz, MobilityLab, APDM Inc., Portland, OR). IMUs were attached at the participant's ankles, and lumbar region using elastic Velcro straps.These sensors are measuring cadence (number of steps taken in 1 minute).
Swing time percent- Physiological measurement of gait | Through study completion, an average of 1 year
  Swing time percent (the percent of time from the total time of one gait cycle that one leg is in the air is measured with the Mobility Lab OPAL system (APDM, USA) consisting of three small inertial measurement units (IMU sensors including 3D accelerometers and 3D gyroscopes sampled at 128 Hz, MobilityLab, APDM Inc., Portland, OR). IMUs were attached at the participant's ankles, and lumbar region using elastic Velcro straps.These sensors are measuring swing time percent (unit are given in percents)
Electrical activity (eeg) of the brain-phisyological measure of electircal signals | Through study completion, an average of 1 year
  During the walking, measure of attention recruitment during walking is applied by a single-channel EEG system (Brain-MARC LTD). The system simplifies EEG analysis to adjust the extraction of relevant attention-related markers from ongoing EEG. EEG is sampled using the MindWave dry electrode system [25], with one frontal electrode (∼Fpz) and one reference electrode on the earlobe. The sampled data are transferred through a wireless connection to the experiment computer, where the signal is processed. An algorithm is calaculating

SECONDARY OUTCOMES:
Cognitive function Go-NoGo Response Inhibition | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically, the Go-NoGo Response Inhibition tests abilities of Attention and Executive Function.
  The Go-NoGo test is a test of response time and response inhibition. Participants are presented with a series of large colored squares at variable delays. Each square may be one of four colors. Participants are instructed to respond as quickly as possible by pressing a mouse button if the square is any color but red. Outcome parameters include accuracy (i.e., percent correct), response time and its associated variance, a composite score computed as accuracy divided by response time, number of errors of omission, number of errors of commission, and response time associated with errors of commission.
Cognitive function-Stroop Interference | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically, Stroop Interference tests abilities of Attention, Executive Function.
  The Stroop test measures response time and executive function. In the test subjects are required to say the color of the word on the screen, not what the word says. Outcome parameters include accuracy, response time and its associated variance, and a composite score computed as accuracy divided by response time.
Cognitive function-Staged Information Processing Speed | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically, Staged Information Processing Speed test abilities of Attention and Information Processing Speed. The Staged Information Processing Speed test measures information processing at increasing levels of complexity. The test is comprised of three levels of information processing load: single digits, two-digit arithmetic problems (e.g., 5-1), and three-digit arithmetic problems (e.g., 3+2-1). Participants are presented with a series of digits or arithmetic problems (as per the level) and are instructed to respond as quickly as possible by pressing the left mouse button if the digit or result is less than or equal to 4 and the right mouse button if it is greater than 4. Outcome parameters for each rate increment for each level include accuracy, response time and its
Cognitive function-Finger Tapping | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically, Finger Tapping tests motor skills. Participants are presented with a white rectangle, which fills with red from left to right over 12 sec. The task requires the participant to tap the left mouse button as many times as possible while the rectangle fills with red. The outcome parameters for this test include inter-tap interval and associated variance (in milliseconds) for the participant's dominant hand.
Cognitive function-'Catch' Game | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically, the 'Catch' Game tests abilities of Executive Function and Motor Skills. During the 'Catch' Game participants see a rectangular white object falling vertically from the top of the screen. Their task is to "catch" the object before it reaches the bottom of the screen by positioning the rectangular green paddle directly in the path of the falling object. Responses are made with the participant's best hand. The rate of the falling object increases incrementally as the test continues making it increasingly difficult to "catch" the object in time. Outcome parameters include response time and associated variance for the first move, number of direction changes per trial, error for missed catches, and a total performance score.
Cognitive function-Problem Solving | Through study completion, an average of 1 year
  NeuroTrax™ computerized tests assess brain wellness across an array of cognitive domains. Specifically,the NeuroTrax Problem Solving test is a non-verbal IQ test that assesses the ability to appreciate the spatial relationships among geometric forms that constitute a pattern. Participants are presented with an incomplete pattern consisting of three squares containing simple geometric forms in a particular configuration. Six additional squares containing geometric forms are presented along the bottom of the screen. Responses with the keyboard number pad indicate which of the six forms best completes the pattern. The spatial relationships among the simple geometric forms become more complex as the test progresses, and the test is adaptive in that it terminates early when performance is poor. The outcome parameter for this test consists of a total accuracy score that incorporates performance at differing levels of difficulty.
Cognitive function-executive function index score | Through study completion, an average of 1 year
  Groups of normalized parameters that measure executive function are averaged to produce index score of executive function. The Outcome Parameters Comprising this Index Scores are: Go-NoGo: Composite Score; Stroop Interference: Composite Score; Catch Game: Total Score.
Cognitive function-Attention index score | Through study completion, an average of 1 year
  Groups of normalized parameters that measure attention are averaged to produce index score of attention. The Outcome Parameters Comprising this Index Scores are: Go-NoGo: Response Time; Go-NoGo: Response Time Standard Deviation; Stroop Interference: Response Time; Staged Info Processing: Response Time; Information Processing: Accuracy.
Cognitive function-Information Processing Speed index score | Through study completion, an average of 1 year
  Groups of normalized parameters that measure Information Processing Speed are averaged to produce index score of Information Processing Speed. The Outcome Parameters Comprising this Index Scores are: Staged Information Processing: Composite Score, Level 1.1; Staged Information Processing: Composite Score, Level 1.3; Staged Information Processing: Composite Score, Level 2.1; Staged Information Processing: Composite Score, Level 2.2
Cognitive function-motor skills index score | Through study completion, an average of 1 year
  Groups of normalized parameters that measure motor skills are averaged to produce index score of motor skills. The Outcome Parameters Comprising this Index Scores are: Finger Tapping: Inter-Tap Interval; Finger Tapping: Tap Interval Std Dev; Catch Game: Time to Make 1st Move

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yogev-Seligmann, Principal Investigator — University of Haifa
Locations (1):
- Galit Yogev-Seligmann, Haifa, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: No